CLINICAL TRIAL: NCT03600168
Title: A Multi-center, Single Arm Post-market Clinical Study to Confirm Safety and Performance of Purastat Absorbable Haemostatic Material for the Management of Bleeding After Open Liver Resection
Brief Title: Post-Market Clinical Study to Confirm Safety and Performance of PuraStat Absorbable Haemostatic Material for the Management of Bleeding in Liver Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: 3-D Matrix Europe SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: PuraStat-001-LIVER
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Liver Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PuraStat® — Synthetic haemostatic material

SUMMARY:
The objective of this post-market clinical follow-up study is to collect medical information on patients implanted with PuraStat®, according to each participating institution's procedures and standards of care.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patient ≥ 18 years old
* Subject have been informed and understand the nature and extent of the study, agree to its provisions and have provided written approved informed consent
* Patient undergoing elective primary or redo open liver resection for hepatic colorectal metastases with a curative intent
* Subject, who, in the opinion of the Clinical Investigator, is able to understand this clinical study, cooperate with the study procedures and is willing to return for the required post-treatment follow-up.

Main Exclusion Criteria:

* Known allergy or hypersensitivity to any component of the investigational treatment PuraStat®
* Pregnant or interested in becoming pregnant during the duration of the study, or breast feeding
* Concurrent participation in another clinical study with a medical device or medicinal product with interfering endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously treated with PuraStat®
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Total Time-To-Haemostasis | Intraoperatively
  Total Time-To-Haemostasis will be intraoperatively measured (minutes, seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- St James' University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No